CLINICAL TRIAL: NCT03341273
Title: Targeted Reduction of Antibiotics Using Procalcitonin in a Multi-center, Randomized, Double-Blinded, Placebo-Controlled Non-Inferiority Study of Azithromycin Treatment in Outpatient Adults With Suspect Lower Respiratory Tract Infection (LRTI) and a Procalcitonin (PCT) Level of < / = 0.25 ng/mL (TRAP-LRTI)
Brief Title: Placebo-Controlled Trial of Antibiotic Therapy in Adults With Suspect Lower Respiratory Tract Infection (LRTI) and a Procalcitonin Level
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to covid
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 15-0020; HHSN272201300015I
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2020-03-12

CONDITIONS: Lower Respiratory Tract Infection
Keywords: Antibiotic Reduction; Antibiotic Therapy; Azyithromycin; Lower Respiratory Tract Infection; Procalcitonin
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Azithromycin (Experimental): 500 mg of Azithromycin (2 capsules of 250 mg) administered orally as a single dose on Day 1, followed by 250 mg capsule of Azithromycin administered orally once daily for 4 days (Day 2 through Day 5). N=337
  Interventions: Drug: Azithromycin; Device: VIDAS B.R.A.H.M.S Procalcitonin Test (PCT)
- Placebo (Placebo Comparator): 2 capsules of Azithromycin placebo administered orally as a single dose on Day 1, followed by 1 capsule of Azithromycin placebo administered orally once daily for 4 days (Day 2 through Day 5). N=337
  Interventions: Other: Placebo; Device: VIDAS B.R.A.H.M.S Procalcitonin Test (PCT)

INTERVENTIONS:
Drug: Azithromycin — Azithromycin is an azalide antibiotic and is derived from erythromycin used to treat many different types of infections caused by bacteria, such as respiratory infections.
  Arms: Azithromycin
Other: Placebo — Placebo will be a matching capsule the same size, weight, and color as the capsules containing Azithromycin tablets.
  Arms: Placebo
Device: VIDAS B.R.A.H.M.S Procalcitonin Test (PCT) — The VIDAS B.R.A.H.M.S PCT is an automated test for use on the VIDAS instruments for the determination of human procalcitonin in human serum or plasma using the Enzyme-Linked Fluorescent Assay (ELFA) technique.

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, non-inferiority multicenter clinical trial of azithromycin vs. placebo in adults presenting as outpatients with suspect Lower Respiratory Tract Infection (LRTI) and a Procalcitonin (PCT) level of < / = 0.25 ng/mL, as a strategy for reducing antibiotic prescriptions. The study is designed to compare the efficacy of azithromycin versus placebo on Day 5 (i.e., after 4 days of treatment) in subjects with suspect LRTI and PCT levels of < / = 0.25 ng/mL at enrollment using a non-inferiority approach. The study will recruit potential subjects 18 years of age or older who are suspected to have LRTI. The enrollment cap will be 840 participants, for the goal of approximately 674 randomized participants who will be randomized 1:1 to receive oral azithromycin or placebo for five days. Randomized subjects will have efficacy measured from the time of the first dose of study drug (Day 1) through approximately Day 28. The Primary Objective is to compare the efficacy of azithromycin versus placebo on Day 5 (i.e., after 4 days of treatment) in subjects with suspect LRTI and PCT levels of < / = 0.25 ng/mL at enrollment using a non-inferiority approach.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, placebo-controlled, non-inferiority multicenter clinical trial of azithromycin vs. placebo in adults presenting as outpatients with suspect Lower Respiratory Tract Infection (LRTI) and a Procalcitonin (PCT) level of < / = 0.25 ng/mL, as a strategy for reducing antibiotic prescriptions. The study is designed to compare the efficacy of azithromycin versus placebo on Day 5 (i.e., after 4 days of treatment) in subjects with suspect LRTI and PCT levels of < / = 0.25 ng/mL at enrollment using a non-inferiority approach. The study will recruit potential subjects 18 years of age or older who are suspected to have LRTI. The enrollment cap will be 840 participants, for the goal of approximately 674 randomized participants who will be randomized 1:1 to receive oral azithromycin or placebo for five days. Randomized subjects will have efficacy measured from the time of the first dose of study drug (Day 1) through approximately Day 28. The primary objective is to compare the efficacy of azithromycin versus placebo on Day 5 (i.e., after 4 days of treatment) in subjects with suspect LRTI and PCT levels of < / = 0.25 ng/mL at enrollment using a non-inferiority approach. The secondary objectives are to compare:1) groups receiving azithromycin versus placebo with regard to all antibiotic use by Days 11 and 28; 2) groups receiving azithromycin versus placebo with regard to return visits to a physician's office or urgent care by Days 11 and 28; 3) groups receiving azithromycin versus placebo with regard to emergency department visits by Days 11 and 28; 4) groups receiving azithromycin versus placebo with regard to hospitalization by Days 11 and 28 if not hospitalized at the enrollment and randomization visit; 5) groups receiving azithromycin versus placebo with regard to improvement in presenting symptoms by Days 11 and 28; 6) the efficacy of azithromycin versus placebo on Day 11 in subjects with suspect LRTI and PCT levels of < / = 0.25 ng/mL at enrollment using a non-inferiority approach; 7) the efficacy of azithromycin versus placebo on Day 28 in subjects with suspect LRTI and PCT levels of < / = 0.25 ng/mL at enrollment using a non-inferiority approach; 8) the efficacy of azithromycin versus placebo in subjects with suspected LRTI and PCT levels of < / = 0.25 ng/mL at Day 5 using a superiority approach, employing the "Response Adjusted for Days of Antibiotic Risk (RADAR)" methodology; 9) groups receiving azithromycin versus placebo in regard to solicited events by Day 5; 10) groups receiving azithromycin versus placebo in regard to hospitalization or visits to an Emergency Department (ED), outpatient clinic, or urgent care center for worsening or persistent LRTI after randomization by Day 5; 11) groups receiving azithromycin versus placebo in regard to improvement in vital sign abnormalities or symptoms present at enrollment, on Day 5; 12) groups receiving azithromycin versus placebo in regard to new vital sign abnormalities or symptoms on Day 5, or deterioration in symptoms relative to the enrollment visit on Day 5.

ELIGIBILITY:
Inclusion Criteria:

1. Clinician suspected Lower Respiratory Tract Infection (LRTI)* based on the presence of at least two qualifying symptoms** OR one qualifying symptom and at least one qualifying vital sign***.

   *LRTI will include acute bronchitis, tracheitis, tracheobronchitis, asthma exacerbation, and acute exacerbation of Chronic obstructive pulmonary disease (COPD) but does not include known pneumonia.

   **New cough, worsening of chronic cough, new sputum production, increased volume or purulence of chronic sputum production, chest pain, and difficulty breathing.

   ***Fever (Provider or patient-measured temperature > / = 37.8 degrees Celsius (100.0 degrees Fahrenheit) or patient-reported feverishness), tachycardia of > / = 90 beats/minute, tachypnea of > 20 breaths/minute.
2. Males and females age > / = 18 years old.
3. Presentation > / = 24 hours and < / = 28 days after the onset of at least one qualifying symptom related to the acute episode of illness.
4. Ability to understand study procedures and willing and able to comply with all required procedures and visits for the entire length of study.
5. Provide written informed consent before initiation of any study procedures.

Exclusion Criteria:

1. Hospitalized prior to screening and enrollment. Subjects enrolled in clinic or Emergency Department (ED) setting and then hospitalized during the same clinical encounter may be included.
2. Chronic pulmonary conditions at the investigator's discretion*.

   *Such as:
   * Noninvasive ventilation use for any indication other than obstructive sleep apnea
   * Long-term invasive mechanical ventilation for any indication
   * Known diagnosis of cystic fibrosis or chronic bronchiectasis.
3. Receipt of an investigational product within 30 days prior to Day 1 or plans to potentially start any investigational product within 30 days after the subject's anticipated study completion.
4. Current enrollment in another clinical trial of an investigational agent.
5. Known or suspected infection at any other anatomic site requiring antibacterial therapy.
6. Immunosuppression*

   *Includes:
   * Human Immunodeficiency Virus (HIV) infection with CD4 < 200 based on last known measurement or patient-reported value
   * History of hematologic malignancies
   * Receipt of chemotherapy within the previous 6 months or anticipated receipt of chemotherapy during the study period (1 month)
   * Known to have an absolute neutrophil count of < 500 cells/mL or an expectation of an absolute neutrophil count of < 500 cells/mL during course of the study
   * Current systemic corticosteroid use (equivalent of 20mg prednisone per day for > / = 2 weeks within the last month)
   * Systemic non-steroid immunosuppressive or biologic therapy for transplant, rheumatologic conditions, or other conditions within the last month. Biologics used specifically for control of moderate to severe asthma, including anti-IgE monoclonal antibody therapy (Xolair) or IL-5 monoclonal antibodies (Mepolizumab and Reslizumab) are allowed
7. Contraindication to the use of azithromycin including history of allergy or intolerance to azithromycin or known prolonged QTc interval (> 500 msec).
8. Any condition that in the judgment of the referring provider or site investigator precludes participation because it could affect subject safety or ability of subject to participate in this trial.
9. Prior use of azithromycin in the past two weeks.
10. Use of any systemic antibiotic in the previous 24 hours.
11. Previous randomization in this trial.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2017-12-08 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-08-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - The Hope Clinic of Emory University, Atlanta, Georgia
  - Atlanta VA Medical Center - Infectious Diseases Clinic, Decatur, Georgia
  - Durham VA Medical Center, Durham, North Carolina
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Texas Medical Center - Michael E. DeBakey Veterans Affairs, Houston, Texas

REFERENCES:
- [Derived] Tsalik EL, Rouphael NG, Sadikot RT, Rodriguez-Barradas MC, McClain MT, Wilkins DM, Woods CW, Swamy GK, Walter EB, El Sahly HM, Keitel WA, Mulligan MJ, Tuyishimire B, Serti E, Hamasaki T, Evans SR, Ghazaryan V, Lee MS, Lautenbach E; TRAP-LRTI Study Group; Antibacterial Resistance Leadership Group. Efficacy and safety of azithromycin versus placebo to treat lower respiratory tract infections associated with low procalcitonin: a randomised, placebo-controlled, double-blind, non-inferiority trial. Lancet Infect Dis. 2023 Apr;23(4):484-495. doi: 10.1016/S1473-3099(22)00735-6. Epub 2022 Dec 13. PMID 36525985

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants, males and non-pregnant females, aged >=18 years, presenting as outpatients with suspected Lower Respiratory Tract Infection (LRTI) with a Procalcitonin (PCT) level of <=0.25 ng/mL were recruited from the community at large. Participants were enrolled between 08DEC2017 and 09MAR2020.
Groups:
- Azithromycin: 500 mg of Azithromycin (2 capsules of 250 mg) administered orally as a single dose on Day 1, followed by 250 mg capsule of Azithromycin administered orally once daily for 4 days (Day 2 through Day 5).
  Azithromycin: Azithromycin is an azalide antibiotic and is derived from erythromycin used to treat many different types of infections caused by bacteria, such as respiratory infections.
  VIDAS B.R.A.H.M.S Procalcitonin Test (PCT): The VIDAS B.R.A.H.M.S PCT is an automated test for use on the VIDAS instruments for the determination of human procalcitonin in human serum or plasma using the Enzyme-Linked Fluorescent Assay (ELFA) technique.
- Placebo: 2 capsules of Azithromycin placebo administered orally as a single dose on Day 1, followed by 1 capsule of Azithromycin placebo administered orally once daily for 4 days (Day 2 through Day 5).
  Placebo: Placebo will be a matching capsule the same size, weight, and color as the capsules containing Azithromycin tablets.
  VIDAS B.R.A.H.M.S Procalcitonin Test (PCT): The VIDAS B.R.A.H.M.S PCT is an automated test for use on the VIDAS instruments for the determination of human procalcitonin in human serum or plasma using the Enzyme-Linked Fluorescent Assay (ELFA) technique.
Period: Overall Study
Arm/Group | Azithromycin | Placebo
Started | 249 | 250
Completed | 229 | 238
Not Completed | 20 | 12
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Enrolled but Treatment Not Administered | 6 | 1
Not completed — Became ineligible after enrollment | 1 | 0
Not completed — Not Eligible at Enrollment | 0 | 1
Not completed — Participant incarcerated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population includes all participants with procalcitonin (PCT) = 0.25 ng/mL who were randomized to receive study product.
Groups:
- Azithromycin: 500 mg of Azithromycin (2 capsules of 250 mg) administered orally as a single dose on Day 1, followed by 250 mg capsule of Azithromycin administered orally once daily for 4 days (Day 2 through Day 5).
- Placebo: 2 capsules of Azithromycin placebo administered orally as a single dose on Day 1, followed by 1 capsule of Azithromycin placebo administered orally once daily for 4 days (Day 2 through Day 5).
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 249 | 250 | 499
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (15.9) | 51.7 (15.0) | 52.2 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 96 | 176
  Male | 169 | 154 | 323
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 16 | 33
  Not Hispanic or Latino | 228 | 233 | 461
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 159 | 146 | 305
  White | 81 | 89 | 170
  More than one race | 2 | 8 | 10
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 249 | 250 | 499

OUTCOME MEASURES:

1. Primary Outcome: Clinical Improvement at Day 5 Visit (D5V)
Description: Clinical improvement at Day 5 Visit is defined as fulfilling all of the following criteria:
  1. Improvement in at least two symptoms present at enrollment or one symptom and at least one vital sign abnormality present at enrollment
  2. Absence of deterioration in any qualifying symptom or new vital sign abnormality not present at enrollment
  3. Absence of fever in the day preceding or at the D5V
  4. No medically attended visit to an ambulatory medical facility or hospitalization for persistent or worsening Lower Respiratory Tract Infection (LRTI) at any time after randomization
Time Frame: Day 5 Visit
Population: The ITT population includes all participants with PCT <= 0.25 ng/mL who were randomized to receive study product.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 249 | 250
percentage of participants | 69 [61 to 77] | 63 [54 to 71]
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Null Hypothesis: Proportion in placebo - Proportion in azithromycin = -12.5%; Test type: Non-Inferiority — The non-inferiority margin is 12.5%. Non-inferiority of placebo is concluded if the lower limit of the 95% confidence interval for the difference in proportions of clinical improvement is greater than -12.5%; The null hypothesis was evaluated using a non-inferiority test and non-inferiority of placebo was concluded if the lower limit of the 95% confidence interval for the difference in proportions of clinical improvement was greater than -12.5%; Risk Difference (RD) = -6, 95% CI 2-sided [-15 to 2] — Multiple imputation with a linear model to impute missing clinical values of improvement. The study day that D5V occurred on was included as a covariate in the final model and the estimates for risk difference assume that study day of D5V is 5

2. Secondary Outcome: Clinical Improvement at Day 11 Visit (D11V)
Description: Clinical improvement at Day 11 Visit is defined as fulfilling all of the following criteria:
  1. Improvement in at least two symptoms present at enrollment or one symptom and at least one vital sign abnormality present at enrollment
  2. Absence of deterioration in any qualifying symptom or new vital sign abnormality not present at enrollment
  3. Absence of fever in the day preceding or at the D11V
  4. No medically attended visit to an ambulatory medical facility or hospitalization for persistent or worsening LRTI at any time after randomization The ITT population includes all participants with PCT = 0.25 ng/mL who were randomized to receive study product.
Time Frame: Day 11 Visit
Population: The ITT population includes all participants with PCT <= 0.25 ng/mL who were randomized to receive study product.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 249 | 250
percentage of participants | 81 [74 to 87] | 76 [70 to 83]
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Null Hypothesis: Proportion in placebo - Proportion in azithromycin = -12.5%; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = -4, 95% CI 2-sided [-12 to 3] — Multiple imputation with a linear model to impute missing clinical values of improvement. The study day that D11V occurred on was included as a covariate in the final model and the estimates for risk difference assume that study day of D11V is 11

3. Secondary Outcome: Clinical Improvement at Day 28 Visit (D28V)
Description: Clinical improvement at Day 28 Visit is defined as fulfilling all of the following criteria:
  1. Improvement in at least two symptoms present at enrollment or one symptom and at least one vital sign abnormality present at enrollment
  2. Absence of deterioration in any qualifying symptom or new vital sign abnormality not present at enrollment
  3. Absence of fever in the day preceding or at the D11V
  4. No medically attended visit to an ambulatory medical facility or hospitalization for persistent or worsening LRTI at any time after randomization
Time Frame: Day 28 Visit
Population: The ITT population includes all participants with PCT <= 0.25 ng/mL who were randomized to receive study product.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 249 | 250
percentage of participants | 88 [83 to 93] | 82 [77 to 86]
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Null Hypothesis: Proportion in placebo - Proportion in azithromycin = -12.5%; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; [p-value comment as in outcome 1, analysis 1]; Risk Difference (RD) = -7, 95% CI 2-sided [-13 to 0] — Multiple imputation with a linear model to impute missing clinical values of improvement. The study day that D11V occurred on was included as a covariate in the final model and the estimates for risk difference assume that study day of D28V is 28

4. Secondary Outcome: Composite Overall Desirability of Outcome Ranking (DOOR) Assessed Employing a Superiority Analysis Using the "Response Adjusted for Days of Antibiotic Risk (RADAR)" Approach at Day 5 Visit
Description: DOOR is a composite endpoint created using clinical outcomes from Day 1 through Day 5 Visit. It is based on adequate clinical improvement at Day 5 Visit and solicited events from Day 1 through Day 5 Visit.
  When comparing two participants with different ordinal clinical outcomes (OCOs), the participant with a better OCO receives a higher DOOR rank. When comparing two participants with the same OCOs, the participant with fewer days of antibiotic use receives a higher DOOR rank.
Time Frame: Day 5 Visit
Population: The ITT population includes all participants with PCT<= 0.25 ng/mL who were randomized to receive study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 249 | 250
Participants
  Adequate clinical improvement (ACI) with no adverse events | 82 | 94
  Adequate clinical improvement with mild adverse events | 47 | 33
  Adequate clinical improvement with moderate adverse events | 25 | 18
  Adequate clinical improvement with severe adverse events | 1 | 3
  No adequate clinical improvement with no medically attended events | 62 | 72
  No ACI with ED, outpatient clinic, or urgent care center visit but no hospitalization | 9 | 15
  No adequate clinical improvement with hospitalization | 1 | 3
  8: Death (any cause) | 0 | 0
  Missing | 22 | 12
Statistical Analysis 1: Comparison: Azithromycin vs Placebo; Null: The sum of the probability that a participant assigned to placebo will have a higher DOOR at Day 5 visit than if assigned to the Azithromycin plus one-half the probability of equal DOORs at Day 5 Visit is 50% (i.e., no difference in DOOR at Day 5 Visit); Test type: Superiority — DOOR is a composite endpoint created using clinical outcomes from Day 1 through Day 5 Visit. It is based on adequate clinical improvement at Day 5 Visit and solicited events from Day 1 through Day 5 Visit; p < 0.001, Wilcoxon (Mann-Whitney) — Missing DOOR values at Day 5 Visit were first imputed using linear regression using baseline covariates and available DOOR components as covariates; The Mann-Whitney test was run on the multiple imputed datasets to generate estimates of DOOR probability and p-value; Pr(Higher DOOR in Placebo at Day 5 Visit = 0.63, 95% CI 2-sided [0.57 to 0.68]

5. Secondary Outcome: Number of Participants Exhibiting Improvement in One or More LRTI Symptoms or Fever at Day 11 Visit
Description: Improvement in LRTI symptoms was defined as presence of at least one-step improvement in the symptom present at baseline. For fever, improvement was defined as changing from presence of fever at baseline to absence of fever at Day 11 Visit.
Time Frame: Day 11 Visit
Population: According-to-protocol at Day 11 (ATP-11) Population includes randomized participants who had no major protocol deviations and consumed 5 doses of study product by D5V, completed their D11V within the protocol defined time window, and had sufficient data to define clinical improvement at D11V.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 211 | 225
Participants | 206 | 221

6. Secondary Outcome: Number of Participants Exhibiting Improvement in One or More LRTI Symptoms or Fever at Day 28 Visit
Description: Improvement in LRTI symptoms was defined as presence of at least one-step improvement in the symptom present at baseline. For fever, improvement was defined as changing from presence of fever at baseline to absence of fever at Day 28 Visit.
Time Frame: Day 28 Visit
Population: ATP-28 Population includes randomized participants who had no major protocol deviations and consumed 5 doses of study product by D5V, completed their D28V within the protocol defined time window, and had sufficient data to define clinical improvement at D28V.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 210 | 223
Participants | 207 | 220

7. Secondary Outcome: Number of Participants Exhibiting Improvement in at Least Two Presenting Signs or Symptoms at Day 5 Visit
Description: Improvement in LRTI symptoms was defined as presence of at least one-step improvement in at least two symptoms present at baseline for participants who qualified based on two symptoms or improvement in one LRTI symptom present at baseline and normalization of one abnormal vital sign at Day 5 Visit for participants who qualified based on one symptom and one vital sign abnormality.
Time Frame: Day 5 Visit
Population: ATP-5 Population includes randomized participants who had no major protocol deviations and consumed 5 doses of study product by D5V, completed their D5V in person within the protocol defined time window, and had sufficient data to define clinical improvement at D5V.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 204 | 221
Participants | 166 | 177

8. Secondary Outcome: Number of Participants Exhibiting Worsening or Deterioration in One or More Symptoms at Day 5 Visit
Description: Clinical deterioration at D5V is defined as at least one-step deterioration (worsening from mild to moderate for example) in any qualifying symptoms or presence of a new vital abnormality at D5V not present at enrollment.
Time Frame: Day 5 Visit
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 204 | 221
Participants | 29 | 32

9. Secondary Outcome: Number of Participants Reporting One or More Hospitalization or Visits to an Emergency Department (ED), Outpatient Clinic, or Urgent Care Center (After Randomization) for Worsening or Persistent Lower Respiratory Tract Infection
Description: This table summarizes the number and percentage of participants reporting any medically attended visits any time after randomization. Note that receipt of a non-study antibiotic after study Day 5 Visit will was not regarded as satisfying this definition if it is related to a new non-respiratory process that is unrelated to the prior diagnosis of LRTI.
Time Frame: Day 1 through Day 5 Visit
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 204 | 221
Participants | 9 | 15

10. Secondary Outcome: Number of Participants Reporting Solicited Adverse Events From Day 1 Through Day 5 Visit
Description: This table summarizes the number and percentage of participants experiencing any solicited events of mild, moderate or severe severity from Day 1 to Day 5 Visit.
Time Frame: Day 1 through Day 5 Visit
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 204 | 221
Participants
  Any Event | 90 | 77
  Abdominal Pain | 47 | 35
  Vomiting | 13 | 10
  Diarrhea | 53 | 55
  Allergic Reaction | 8 | 9
  Candidiasis | 8 | 8

11. Secondary Outcome: Number of Participants With One or More Emergency Department Visits for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) by Day 11 Visit
Description: This table summarizes the number of participants with one or more Emergency Department Visits for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) from Day 1 through Day 11 Visit.
Time Frame: Day 1 through Day 11
Population: ATP-11 Population includes randomized participants who had no major protocol deviations and consumed 5 doses of study product by D5V, completed their D11V within the protocol defined time window, and had sufficient data to define clinical improvement at D11V.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 221 | 225
Participants | 3 | 9

12. Secondary Outcome: Number of Participants With One or More Emergency Department Visits for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) by Day 28 Visit
Description: This table summarizes the number of participants with one or more Emergency Department Visits for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) in Azithromycin Group from Day 1 through Day 28 Visit.
Time Frame: Day 1 through Day 28 Visit
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 210 | 223
Participants | 3 | 9

13. Secondary Outcome: Number of Participants With One or More Hospitalizations (if Not Hospitalized at Enrollment) for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) by Day 11 Visit
Description: This table summarizes the number of participants with one or more hospitalizations for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) from Day 1 through Day 11 Visit.
Time Frame: Day 1 through Day 11 Visit
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 211 | 225
Participants | 1 | 1

14. Secondary Outcome: Number of Participants With One or More Hospitalizations (if Not Hospitalized at Enrollment) for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) by Day 28 Visit
Description: This table summarizes the number of participants with one or more hospitalizations for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) from Day 1 through Day 28 Visit.
Time Frame: Day 1 through Day 28 Visit
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 210 | 223
Participants | 1 | 1

15. Secondary Outcome: Number of Participants With One or More Unplanned Return to a Physician's Office or Urgent Care for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) by Day 11 Visit
Description: This table summarizes the number of participants with one or more unplanned Return to a Physician's Office or Urgent Care for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) from Day 1 through Day 11 Visit.
Time Frame: Day 1 through Day 11 Visit
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 211 | 225
Participants | 5 | 7

16. Secondary Outcome: Number of Participants With One or More Unplanned Return to a Physician's Office or Urgent Care for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) by Day 28 Visit
Description: This table summarizes the number of participants with one or more unplanned Return to a Physician's Office or Urgent Care for Persistent or Worsening Lower Respiratory Tract Infection (LRTI) from Day 1 through Day 28 Visit.
Time Frame: Day 1 through Day 28 Visit
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 210 | 223
Participants | 6 | 7

17. Secondary Outcome: Number of Participants With a New Occurrence of a Vital Sign Abnormality at Day 5 Visit
Description: This table summarizes the number and percentage of participants experiencing new vital signs abnormalities at Day 5 Visit that were not present at baseline.
Time Frame: Day 5 Visit
Population: ATP-5 Population includes randomized participants who had no major protocol deviations and consumed 5 doses of study product by D5V, completed their D5V in person within the protocol defined time window, and had sufficient data to define clinical improvement at D5V. For vital signs, only participants with without the vital sign abnormality are analyzed. For fever, only participants with non-missing values for fever are analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 202 | 216
Participants
  Any Vital Sign | 19 | 24
  Temperature | 0 | 0
  Pulse: number analyzed (Participants) | 142 | 128
  Pulse | 17 | 19
  Respiratory Rate: number analyzed (Participants) | 189 | 197
  Respiratory Rate | 3 | 5

18. Secondary Outcome: Quantification of All Antibiotic Use From Day 1 Through Day 11 Visit
Description: The table summarizes the mean number of days of antibiotic use including study and non-study antibiotics for participants from Day 1 through Day 11 Visit.
Time Frame: Day 1 through Day 11 Visit
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 211 | 225
days | 5.1 [5.0 to 5.3] | 0.3 [0.1 to 0.5]

19. Secondary Outcome: Quantification of All Antibiotic Use From Day 1 Through Day 28 Visit
Description: The table summarizes the mean number of days of antibiotic use including study and non-study antibiotics for participants from Day 1 through Day 28 Visit.
Time Frame: Day 1 through Day 28 Visit
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 210 | 223
days | 5.5 [5.2 to 5.9] | 0.9 [0.5 to 1.4]

ADVERSE EVENTS:
Time Frame: Solicited Adverse Events were collected from Day 1 through Day 11. As the safety profile of azithromycin is well established, and this trial was not powered to detect new, unknown safety signals, there was no azithromycin-related Adverse Event (AE) collection or Serious Adverse Events (SAEs) reporting during this study. Unanticipated adverse device effect (UADE) were unexpected, but were to be reported appropriately if they occurred during the study.
Description: Serious adverse events were not collected for this study, therefore the number of participants at risk for serious adverse events is zero.
Arm/Group | Azithromycin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/242 | 0/247
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 114/242 | 97/247
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=242) | Placebo (N=247)
Abdominal Pain (Gastrointestinal disorders) | 61 (160) | 43 (119)
Diarrhoea (Gastrointestinal disorders) | 73 (232) | 65 (229)
Vomiting (Gastrointestinal disorders) | 16 (30) | 16 (33)
Candida Infection (Infections and infestations) | 14 (59) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT03341273/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/73/NCT03341273/SAP_001.pdf